CLINICAL TRIAL: NCT05983042
Title: Effect of CYP2C9*3 rs 1057910 Polymorphism on the Efficacy and Tolerability of Ibuprofen After Molar Tooth Extraction in Pakistani Population
Brief Title: Effect of CYP2C9*3 Polymorphism on Ibuprofen in Pakistani Population
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: Riphah/IIMC/IRC/22/2072
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood was withdrawn, and DNA extraction was performed using Chelex method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Ibuprofen — Ibuprofen 400mg three times a day for three days

SUMMARY:
The goal of this Observational study was to identify the effect of CYP2C9 gene polymorphism in the Pakistani population. The main question it aims to answer were:

* to evaluate the effect of this genetic polymorphism on the clinical efficacy of Ibuprofen
* to evaluate the effect of this genetic polymorphism on the clinical tolerability of Ibuprofen Participants were prescribed Ibuprofen after molar tooth extraction.

DETAILED DESCRIPTION:
The goal of this observational study was to identify the effect of CYP2C9*3 gene polymorphism in the Pakistani population, due to the high prevalence of this variant in the Pakistani Population

The main question it aims to answer were:

* to evaluate the effect of this genetic polymorphism on the clinical efficacy of Ibuprofen
* to evaluate the effect of this genetic polymorphism on the clinical tolerability of Ibuprofen Participants were prescribed Ibuprofen after molar tooth extraction.

The blood samples of the participants were taken and further genotyping was performed using conventional tetraARMS PCR. The results were visualized by gel electrophoresis.

ELIGIBILITY:
Inclusion Criteria:

* Pakistani individuals
* Absence of systemic diseases
* Extractions required based on orthodontic, periodontal, and endodontic indications

Exclusion Criteria:

* history of bleeding or gastrointestinal ulcers
* allergic to ibuprofen or other NSAIDs.
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals who were advised for molar tooth extractions based on orthodontic, periodontal, and endodontic indications
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the genetic variabilities in the clinical efficacy of ibuprofen after molar tooth extraction using a visual analog scale VAS | three days
  A Visual Analogue Scale (VAS) is one of the self-administered pain rating scales, to measure pain intensity. The pain was interpreted as no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).

SECONDARY OUTCOMES:
To evaluate the genetic variabilities in the tolerability of ibuprofen after molar tooth extraction using the General Assessment of Side Effects GASE scale. | three days
  The self-rating scale General Assessment of Side Effects (GASE), is about the most frequent side effects in clinical trials of different drugs. Every symptom (dyspepsia, nausea, diarrhea) had to be answered twice: first, participants had to rate the intensity of this symptom during the last 3 days, and second, if this symptom was present, participants had to rate whether they attribute it to current drug intake.

CONTACTS AND LOCATIONS:
Overall Officials: Ammarah Amjad, BDS, Principal Investigator — Riphah International University
Locations (1):
- Ammarah Amjad, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No